CLINICAL TRIAL: NCT02376244
Title: A Randomised Controlled Trial on the Efficacy of High Intensity Interval Training Compared With Moderate Intensity Interval Training for Patients Undergoing Cardiac Rehabilitation
Brief Title: The Health Impact of High Intensity Exercise Training With Intervals During Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP 006 - HIIT
Record Dates: First submitted 2015-02-11; First posted 2015-03-03 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Heart Disease; Heart Attacks
Keywords: High intensity Interval Exercise training; Cardiac rehabilitation; cardiac revascularisation; Percutaneous coronary interventions; Cardiac surgery
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction | interventions — High-Intensity Interval Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity interval training (HIIT) (Experimental): Patients will undergo a 15-minute warm-up, followed by a 24-minute conditioning phase, and a 10-minute cool-down. The conditioning phase will include a combination of aerobic exercise (e.g. cycling or walking) and resistance exercise (e.g. squats, bicep curls). Patients will complete 5 intervals of 3 minutes with 2 minute rest periods interspersed. The intensity will correspond to 16-17 on the Borg 6-20 Rating of perceived exertion scale.
  Patients will exercise once a week for 8 weeks.
  Interventions: Other: High intensity interval training (HIIT)
- Standard Care (Active Comparator): Patients assigned to this group will participate in usual standard care of cardiac rehabilitation.
  Commonly, patients will undergo a 15-minute warm-up, followed by a 24-minute conditioning phase, and a 10-minute cool-down. The conditioning phase will include a combination of aerobic exercise (e.g. cycling or walking) and resistance exercise (e.g. squats, bicep curls). Patients will complete 5 intervals of 3 minutes with 2 minute rest periods interspersed. The intensity will correspond to 11-15 on the Borg 6-20 Rating of perceived exertion scale.
  Patients will exercise once a week for 8 weeks.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: High intensity interval training (HIIT) — Standard care cardiac rehabilitation classes, delivered at a higher exercise intensity
  Other Names: Group 1
  Arms: High intensity interval training (HIIT)
Other: Standard care — Standard care cardiac rehabilitation according to current guidelines
  Other Names: Group 2
  Arms: Standard Care

SUMMARY:
Cardiac rehabilitation is a program designed to help patients regain good health through lifestyle change after a heart attack, heart surgery or other heart problems. Patients will take part in exercise sessions and education lessons, tailored to meet their personal needs. The exercise training component of cardiac rehabilitation may be delivered as intervals of short intense sessions (also known as high intensity intervals) or the current standard care of longer but less intense sessions (moderate intense intervals). Both exercises have been shown to increase fitness levels and also prevent future risk of heart disease.

The purpose of this study is to determine the efficacy and safety of high intensity interval exercise training (HIIT) in patients who had a recent cardiac revascularization procedure or recovering from a heart attack, in comparison to current standard of moderate intensity exercise training in terms of their physical fitness and psychological well-being.

DETAILED DESCRIPTION:
Cardiac rehabilitation is an eight week program designed to help patients regain good health through changed lifestyle after a possible heart attack, heart surgery or other heart problems. Patients will take part in exercise sessions and education lessons, tailored to meet their personal needs. The exercise training component of cardiac rehabilitation may be delivered as intervals of short intense sessions (also known as high intensity intervals) or the current standard care of longer but less intense sessions (moderate intense intervals). Both exercises have been shown to increase fitness levels and also prevent future risk of heart disease. Although there is some evidence to suggest that high intensity interval training produces better body muscles recovery and fitness during cardiac rehabilitation, many important health outcomes have not yet been determined. Such outcomes include the ability of the body to safely control blood pressure and heartbeat rate. Others include health-related quality of life and emotional well-being.

This study will explore whether there are any differences in health outcomes before and after the introduction of the intervention for patients undergoing high intensity interval exercise compared to those on moderate intensity interval exercise in terms of the recovery of the ability to control blood pressure and heartbeat rate, and also health-related quality of life and emotional well-being. In addition, patients' opinions will be sought regarding pain levels, the acceptability and the extent of enjoyment they get from each of the two types of exercise training.

For each patient, their exercise program will be designed to match their preferences and requirements. Some may prefer to work in a gym environment and so will have their program designed around this type of activity. Others may prefer to work in a group exercise circuit, with their program matched to what is available. When comparing the two types of exercise, everything will be kept the same; from the warm up and cool down, to the types of movements; the only thing that will change is the intensity of the exercise.

Before and after the eight week training program, patients will be asked to have an assessment to measure the effects that the exercise has on their body. Things like heart rate and blood pressure will be taken and they will also undergo a physical fitness test.

After the training, patients will complete questionnaires to establish their level of enjoyment of the program, how motivated they were to complete it. In addition, their quality of life and emotional well-being will be measured by completing questionnaires before and after the 8 weeks of the cardiac rehabilitation program. The investigators anticipate that a total of 46 patients will be recruited for the study over a period of 6 months. In the United Kingdom, it is believed that delivering an improved exercise training program has the potential to enhance patients' recovery from heart disease that may reduce the need for hospital services and therefore a better use of the National Health Service resources.

ELIGIBILITY:
Inclusion Criteria:

* History of acute coronary syndromes, had a recent revascularization procedure
* History of stable heart failure or stable angina.

Exclusion Criteria:

* Unstable angina
* Systolic blood pressure of >200 mm Hg, or diastolic blood pressure >110 mm Hg (should be assessed on a case-by-case basis)
* Orthostatic blood pressure drop of >20 mm Hg with symptoms
* May have had the implantation of cardiac defibrillators (ICD)
* Synchronization devices or ventricular assist devices
* Have had a heart valve repair/replacement, a heart transplant, or grown-up congenital heart disease, critical aortic stenosis, acute systemic illness or fever, -
* Uncontrolled atrial or ventricular arrhythmias, acute pericarditis or myocarditis
* Recent embolism, thrombophlebitis, resting S-T segment depression (>2 mm), uncontrolled diabetes (should be assessed in accordance with local protocol and on a case-by-case basis)
* Severe orthopedic conditions that would prohibit exercise
* Other metabolic conditions, such as acute thyroiditis, hypokalemia or hyperkalemia, hypovolemia, severe rejection (cardiac transplant recipients), triple A >4.5 cm (if under surveillance will need confirmation from vascular surgeon as long as blood pressure remains stable)
* Tachycardia >100 beats per minute at rest, or cataracts (may commence exercise after 6 weeks)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in Heart Rate Variability (as measured by a hemodynamic monitoring system) | Change from baseline in heart rate variability at 8 weeks after the start of the intervention
  The primary outcome is the difference in heart rate variability between baseline and 8 weeks after the start of the intervention measured using finger photoplethysmography

SECONDARY OUTCOMES:
Changes in Baroreflex Sensitivity (as measured by a hemodynamic monitoring system) | Change from baseline in baroreflex sensitivity at 8 weeks after the start of the intervention
  This is the difference in heart rate variability between baseline and 8 weeks after the start of intervention measured using finger photoplethysmography
Changes in Peak Oxygen Uptake (as measured by a submaximal exercise test) | Changes in peak oxygen uptake between baseline and 8 weeks after the start of intervention
  Submaximal Cardiopulmonary Exercise Testing will be performed to measure changes in peak oxygen uptake between baseline and 8 weeks after the start of the intervention
Changes in Enjoyment of Exercise (as measured by a questionnaire) | Changes in perception of enjoyment of exercise at between baseline and 8 weeks after the start of intervention
  Changes in pleasure and displeasure, affect, arousal between baseline and 8 weeks after the start of intervention will be assessed by using a "Feelings Scale", "Felt Arousal Scale", "Physical Activity Enjoyment Scale" respectively.
Changes in health-related Quality of Life (as measured by a questionnaire) | Changes in health-related quality of life between baseline and 8 weeks after the start of intervention
  Changes in health-related quality of life between baseline and 8 weeks after the start of intervention will be measured by completion of MacNew Quality of Life questionnaires
Changes in Rating of Perceived Exertion (as measured by a scale) | Changes in the rating of perceived exertion between baseline and 8 weeks after start of intervention
  Ratings of perceived exertion (RPE) allow the intensity of exercise to be determined subjectively on a scale of 6-20. Changes in RPE scales will be assessed at start of each workout as part of service protocol to gauge patient effort, fatigue and muscular discomfort and the differences between baseline and 8 weeks after start of intervention will be determined. At the end of each session, patients will be expected to submit an overall session RPE of how they perceived the entire exercise session (Kilpatrick et al. 2014).

OTHER OUTCOMES:
Changes in reported incidents of acute pain (as measured by a visual analogue scale) | Changes between baseline incidents of acute pain and 8 weeks after start of intervention
  Pain is a contributing factor to the displeasure experienced during some exercise (Ekkekakis et al. 2012). For this reason participants will be required to complete a visual analogue scale to quantify any pain during the sessions. Changes in perception of pain will assessed between baseline and 8 weeks after the start of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alison C Welsh, Principal Investigator — Edge Hill University and Liverpool Heart and Chest Hospital; Adrian Roose, Principal Investigator — Liverpool Heart and Chest Hospital; Joseph Mills, Principal Investigator — Liverpool Heart and Chest Hospital; Bashir Matata, Principal Investigator — Liverpool Heart and Chest Hospital; Adrian Midgley, Principal Investigator — Edge Hill University; Felipe Cunha, Principal Investigator — Edge Hill University
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munk PS, Butt N, Larsen AI. High-intensity interval exercise training improves heart rate variability in patients following percutaneous coronary intervention for angina pectoris. Int J Cardiol. 2010 Nov 19;145(2):312-314. doi: 10.1016/j.ijcard.2009.11.015. Epub 2009 Dec 5. PMID 19962772
- [Result] Guiraud T, Nigam A, Gremeaux V, Meyer P, Juneau M, Bosquet L. High-intensity interval training in cardiac rehabilitation. Sports Med. 2012 Jul 1;42(7):587-605. doi: 10.2165/11631910-000000000-00000. PMID 22694349
- [Result] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Result] Currie KD, Rosen LM, Millar PJ, McKelvie RS, MacDonald MJ. Heart rate recovery and heart rate variability are unchanged in patients with coronary artery disease following 12 weeks of high-intensity interval and moderate-intensity endurance exercise training. Appl Physiol Nutr Metab. 2013 Jun;38(6):644-50. doi: 10.1139/apnm-2012-0354. Epub 2013 Jan 17. PMID 23724882